CLINICAL TRIAL: NCT03510884
Title: A Randomized, Double-Blind, Placebo-Controlled Study Followed by an Open Label Treatment Period to Evaluate the Efficacy and Safety of Alirocumab in Children and Adolescents With Heterozygous Familial Hypercholesterolemia
Brief Title: An Efficacy and Safety Study of Alirocumab in Children and Adolescents With Heterozygous Familial Hypercholesterolemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EFC14643; 2017-001903-60 (EudraCT Number); U1111-1193-0721 (Other: UTN)
Record Dates: First submitted 2018-04-18; First posted 2018-04-27 (Actual); Results first posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Hypercholesterolaemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — alirocumab; Rosuvastatin Calcium; Atorvastatin; Simvastatin; Pravastatin; Lovastatin; Fluvastatin; Ezetimibe; Cholestyramine Resin; Niacin; Fenofibrate; Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo/Alirocumab Q2W (Experimental): Participants received subcutaneous (SC) injection of placebo (matched to alirocumab) based on their body weight (BW) (less than [<] 50 kilograms [kg] or greater than or equal to [>=] 50 kg) Q2W for 24 weeks in DB treatment period added to stable LMT. After completion of DB treatment period, eligible participants entered into OL treatment period and received alirocumab 40 milligrams (mg) (for BW <50 kg) or 75 mg (for BW >=50 kg) Q2W from Week 24 up to an additional 80 weeks (i.e., up to Week 104) added to stable LMT. After Week 24, dose up-titrated from 40 mg to 75 mg when BW increased from <50 kg to >=50 kg. From Week 32 up to Week 104, based on participant LDL-C value, alirocumab dose was either up-titrated as 40 mg to 75 mg (for BW <50 kg) or 75 mg to 150 mg (for BW >=50 kg) or down titrated as 75 mg to 40 mg (for BW <50 kg) or 150 mg to 75 mg (for BW >=50 kg).
  Interventions: Drug: Alirocumab SAR236553 (REGN727); Drug: Rosuvastatin; Drug: Atorvastatin; Drug: Simvastatin; Drug: Pravastatin; Drug: Lovastatin; Drug: Fluvastatin; Drug: Ezetimibe; Drug: Cholestyramine; Drug: Nicotinic acid; Drug: Fenofibrate; Drug: Omega-3 fatty acids; Drug: Placebo
- Alirocumab Q2W (Experimental): Participants received SC injection of alirocumab 40 mg (for BW <50 kg) or 75 mg (for BW >=50 kg) Q2W for 24 weeks in DB treatment period added to stable LMT. Alirocumab dose was up-titrated to 75 mg or 150 mg Q2W from Week 12, when LDL-C level was >=110 milligrams per deciliter (mg/dL) (2.85 millimoles per liter [mmol/L]) at Week 8. After completion of DB treatment period, eligible participants entered into OL treatment period and received alirocumab 40 mg (for BW <50 kg) or 75 mg (for BW >=50 kg) from Week 24 up to an additional 80 weeks (i.e., up to Week 104) added to stable LMT. After Week 24, dose up-titrated from 40 mg to 75 mg when BW increased from <50 kg to >=50 kg. From Week 32 up to Week 104, based on participant LDL-C value, alirocumab dose was either up-titrated as 40 mg to 75 mg (for BW <50 kg) or 75 mg to 150 mg (for BW >=50 kg) or down titrated as 75 mg to 40 mg (for BW <50 kg) or 150 mg to 75 mg (for BW >=50 kg).
  Interventions: Drug: Alirocumab SAR236553 (REGN727); Drug: Rosuvastatin; Drug: Atorvastatin; Drug: Simvastatin; Drug: Pravastatin; Drug: Lovastatin; Drug: Fluvastatin; Drug: Ezetimibe; Drug: Cholestyramine; Drug: Nicotinic acid; Drug: Fenofibrate; Drug: Omega-3 fatty acids
- Placebo/Alirocumab Q4W (Experimental): Participants received SC injection of placebo (matched to alirocumab) based on their BW (<50 kg or >=50 kg) Q4W for 24 weeks in DB treatment period added to stable LMT. After completion of DB treatment period, eligible participants entered into OL treatment period and received alirocumab 150 mg (for BW <50 kg) or 300 mg (for BW >=50 kg) Q4W from Week 24 up to an additional 80 weeks (i.e., up to Week 104) added to stable LMT. After Week 24, dose up-titrated from 150 mg to 300 mg when BW increased from <50 kg to >=50 kg. From Week 32 up to Week 104, based on participant LDL-C value, alirocumab dose was either up-titrated as 150 mg Q4W to 75 mg Q2W (for BW <50 kg) or 300 mg Q4W to 150 mg Q2W (for BW >=50 kg) or down titrated as 75 mg Q2W to 40 mg Q2W (for BW <50 kg) or 150 mg Q2W to 75 mg Q2W (for BW >=50 kg).
  Interventions: Drug: Alirocumab SAR236553 (REGN727); Drug: Rosuvastatin; Drug: Atorvastatin; Drug: Simvastatin; Drug: Pravastatin; Drug: Lovastatin; Drug: Fluvastatin; Drug: Ezetimibe; Drug: Cholestyramine; Drug: Nicotinic acid; Drug: Fenofibrate; Drug: Omega-3 fatty acids; Drug: Placebo
- Alirocumab Q4W (Experimental): Participants received SC injection of alirocumab 150 mg (for BW <50 kg) or 300 mg (for BW >=50 kg) Q4W for 24 weeks in DB treatment period added to stable LMT. Alirocumab dose was up-titrated to 75 mg or 150 mg Q2W from Week 12, when LDL-C level >=110 mg/dL (2.85 mmol/L) at Week 8. After completion of DB treatment period, eligible participants entered into OL treatment period and received alirocumab 150 mg (for BW <50 kg) or 300 mg (for BW >=50 kg) from Week 24 up to an additional 80 weeks (i.e., up to Week 104) added to stable LMT. After Week 24, dose up-titrated from 150 mg to 300 mg when BW increased from <50 kg to >=50 kg. From Week 32 up to Week 104, based on participant LDL-C value, alirocumab dose was either up-titrated as 150 mg Q4W to 75 mg Q2W (for BW <50 kg) or 300 mg Q4W to 150 mg Q2W (for BW >=50 kg) or down titrated as 75 mg Q2W to 40 mg Q2W (for BW <50 kg) or 150 mg Q2W to 75 mg Q2W (for BW >=50 kg).
  Interventions: Drug: Alirocumab SAR236553 (REGN727); Drug: Rosuvastatin; Drug: Atorvastatin; Drug: Simvastatin; Drug: Pravastatin; Drug: Lovastatin; Drug: Fluvastatin; Drug: Ezetimibe; Drug: Cholestyramine; Drug: Nicotinic acid; Drug: Fenofibrate; Drug: Omega-3 fatty acids

INTERVENTIONS:
Drug: Alirocumab SAR236553 (REGN727) — Pharmaceutical form:solution Route of administration: subcutaneous injection
  Other Names: Praluent
Drug: Rosuvastatin — Pharmaceutical form:tablet Route of administration: oral
Drug: Atorvastatin — Pharmaceutical form:Tablet Route of administration: Oral
Drug: Simvastatin — Pharmaceutical form:Tablet Route of administration: Oral
Drug: Pravastatin — Pharmaceutical form:Tablet Route of administration: Oral
Drug: Lovastatin — Pharmaceutical form:Tablet Route of administration: Oral
Drug: Fluvastatin — Pharmaceutical form:Capsule Route of administration: Oral
Drug: Ezetimibe — Pharmaceutical form:Tablet Route of administration: Oral
Drug: Cholestyramine — Pharmaceutical form:oral suspension Route of administration: oral
Drug: Nicotinic acid — Pharmaceutical form:Tablet Route of administration: Oral
Drug: Fenofibrate — Pharmaceutical form:Tablet Route of administration: Oral
Drug: Omega-3 fatty acids — Pharmaceutical form:capsule Route of administration: oral
Drug: Placebo — Pharmaceutical form:solution Route of administration: subcutaneous injection
  Arms: Placebo/Alirocumab Q2W; Placebo/Alirocumab Q4W

SUMMARY:
Primary Objective:

To evaluate the efficacy of alirocumab administered every 2 weeks (Q2W) and every 4 weeks (Q4W) versus placebo after 24 weeks of double-blind (DB) treatment on low-density lipoprotein cholesterol (LDL-C) levels in participants with heterozygous familial hypercholesterolemia (heFH) 8 to 17 years of age on optimal stable daily dose of statin therapy ± other lipid modifying therapies (LMTs) or a stable dose of non-statin LMTs in case of intolerance to statins.

Secondary Objectives:

* To evaluate the efficacy of alirocumab versus placebo on LDL-C levels.
* To evaluate the effects of alirocumab versus placebo on other lipid parameters.
* To evaluate the safety and tolerability of alirocumab in comparison with placebo.
* To evaluate the efficacy, safety, and tolerability of alirocumab after open label treatment.
* To evaluate the development of anti-alirocumab antibodies.

DETAILED DESCRIPTION:
The study duration was approximately up to 110 weeks (run-in period [if needed]: up to 4 weeks [+2 days], screening period: up to 2 weeks [+5 days], double-blind treatment period: 24 weeks, open label (OL) treatment period: 80 weeks).

ELIGIBILITY:
Inclusion criteria:

* Children and adolescent male and female participants 8 to 17 years of age at the time of signed informed consent.
* Participants with diagnosis of heFH through genotyping or clinical criteria.
* Participants treated with optimal dose of statin +/- other LMT(s) or non-statin LMT(s) if statin intolerant at stable dose for at least 4 weeks prior to screening lipid sampling.
* Participants with calculated LDL-C greater than or equal to 130 mg/dL (>=3.37 mmol/L) at the screening visit except for participants who have previously participated in the DFI14223 (NCT02890992) study.
* A signed informed consent indicating parental permission with or without participant assent.

Exclusion criteria:

* Participant with body weight < 25 kg.
* Participants aged of 8 to 9 years not at Tanner stage 1 and participants aged of 10 to 17 years not at least at Tanner stage 2 in their development.
* Participants with secondary hyperlipidemia.
* Diagnosis of homozygous familial hypercholesterolemia.
* Participant who had received lipid apheresis treatment within 2 months prior to the screening period, or has plans to receive it during the study.
* Participants with uncontrolled type 1 or type 2 diabetes mellitus.
* Participants with known uncontrolled thyroid disease.
* Participants with uncontrolled hypertension.
* Fasting triglycerides greater than (>) 350 mg/dL (3.95 mmol/L).
* Severe renal impairment (ie, estimated glomerular filtration rate <30 mL/min/1.73 m^2).
* Alanine aminotransferase or aspartate aminotransferase >2*upper limit of normal (ULN).
* Creatinine phosphokinase (CPK) >3*ULN.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 153 (Actual)
Dates: Start 2018-05-31 (Actual); Primary Completion 2021-01-14 (Actual); Study Completion 2022-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (43):
- United States (5):
  - Excel Medical Clinical Trials, LLC-Site Number:8400001, Boca Raton, Florida
  - Washington University School of Medicine-Site Number:8400006, St Louis, Missouri
  - Presbyterian Novant Heart & Wellness-Site Number:8400002, Charlotte, North Carolina
  - Cincinnati Children's Hospital Medical Center-Site Number:8400005, Cincinnati, Ohio
  - Vanderbilt University-Site Number:8400003, Nashville, Tennessee
- Investigational Site Number :0320001, Buenos Aires, Argentina
- Investigational Site Number :0400001, Vienna, Austria
- Brazil (2):
  - Investigational Site Number :0760004, Porto Alegre, Rio Grande do Sul
  - Investigational Site Number :0760001, São Paulo
- Investigational Site Number :1000002, Plovdiv, Bulgaria
- Investigational Site Number :1240001, Québec, Canada
- Czechia (2):
  - Investigational Site Number :2030002, Brno
  - Investigational Site Number :2030001, Praha 5 - Motol
- Investigational Site Number :2080001, Copenhagen, Denmark
- Investigational Site Number :2460001, HUS, Finland
- France (2):
  - Investigational Site Number :2500001, Bron
  - Investigational Site Number :2500002, Nantes
- Investigational Site Number :3480001, Budapest, Hungary
- Italy (3):
  - Investigational Site Number :3800003, Milan
  - Investigational Site Number :3800001, Palermo
  - Investigational Site Number :3800002, Roma
- Lebanon (2):
  - Investigational Site Number :4220001, Beirut
  - Investigational Site Number :4220003, Room Hospital Street, Achrafie
- Mexico (2):
  - Investigational Site Number :4840008, Guadalajara, Jalisco
  - Investigational Site Number :4840007, Oaxaca City
- Investigational Site Number :5280001, Amsterdam, Netherlands
- Investigational Site Number :5780001, Oslo, Norway
- Poland (2):
  - Investigational Site Number :6160002, Gdansk, Pomeranian Voivodeship
  - Investigational Site Number :6160001, Lodz
- Russia (4):
  - Investigational Site Number :6430006, Kazan'
  - Investigational Site Number :6430001, Kemerovo
  - Investigational Site Number :6430004, Moscow
  - Investigational Site Number :6430002, Ufa
- Investigational Site Number :7050001, Ljubljana, Slovenia
- Investigational Site Number :7100002, Parow, South Africa
- Spain (4):
  - Investigational Site Number :7240003, Pamplona, Navarre
  - Investigational Site Number :7240002, A Coruña
  - Investigational Site Number :7240004, Badalona
  - Investigational Site Number :7240001, Barcelona
- Investigational Site Number :7520001, Stockholm, Sweden
- Investigational Site Number :1580001, Taipei, Taiwan
- Turkey (Türkiye) (2):
  - Investigational Site Number :7920002, Ankara
  - Investigational Site Number :7920001, Izmir

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Santos RD, Wiegman A, Caprio S, Cariou B, Averna M, Poulouin Y, Scemama M, Manvelian G, Garon G, Daniels S. Alirocumab in Pediatric Patients With Heterozygous Familial Hypercholesterolemia: A Randomized Clinical Trial. JAMA Pediatr. 2024 Mar 1;178(3):283-293. doi: 10.1001/jamapediatrics.2023.6477. PMID 38315470

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 43 active sites in 24 countries. A total of 203 participants were screened between 31-May-2018 and 31-Jul-2020, of whom 50 were screen failures. Screen failures were mainly due to exclusion criteria met. A total of 153 participants were randomized with a 2:1 ratio to receive study treatment (alirocumab: placebo).
Pre-assignment Details: Randomization was stratified according to previous participation (yes or no) in the Phase 2 DFI14223 (NCT02890992) study and Baseline body weight (BW) (less than [<] 50 kilograms (kg) or greater than or equal to [>=] 50 kg).
Groups:
- Placebo/Alirocumab Q2W: Participants received subcutaneous (SC) injection of placebo (matched to alirocumab) based on their BW (<50 kg or >=50 kg) every 2 weeks (Q2W) for 24 weeks in double-blind (DB) treatment period added to stable lipid modifying therapy (LMT). After completion of DB treatment period, eligible participants entered into open-label (OL) treatment period and received alirocumab 40 milligrams (mg) (for BW <50 kg) or 75 mg (for BW >=50 kg) Q2W from Week 24 up to an additional 80 weeks (i.e., up to Week 104) added to stable LMT. After Week 24, dose up-titrated from 40 mg to 75 mg when BW increased from <50 kg to >=50 kg. From Week 32 up to Week 104, based on participant low density lipoprotein cholesterol (LDL-C) value, alirocumab dose was either up-titrated as 40 mg to 75 mg (for BW <50 kg) or 75 mg to 150 mg (for BW >=50 kg) or down titrated as 75 mg to 40 mg (for BW <50 kg) or 150 mg to 75 mg (for BW >=50 kg).
- Placebo/Alirocumab Q4W: Participants received SC injection of placebo (matched to alirocumab) based on their BW (<50 kg or >=50 kg) every 4 weeks (Q4W) for 24 weeks in DB treatment period added to stable LMT. After completion of DB treatment period, eligible participants entered into OL treatment period and received alirocumab 150 mg (for BW <50 kg) or 300 mg (for BW >=50 kg) Q4W from Week 24 up to an additional 80 weeks (i.e., up to Week 104) added to stable LMT. After Week 24, dose up-titrated from 150 mg to 300 mg when BW increased from <50 kg to >=50 kg. From Week 32 up to Week 104, based on participant LDL-C value, alirocumab dose was either up-titrated as 150 mg Q4W to 75 mg Q2W (for BW <50 kg) or 300 mg Q4W to 150 mg Q2W (for BW >=50 kg) or down titrated as 75 mg Q2W to 40 mg Q2W (for BW <50 kg) or 150 mg Q2W to 75 mg Q2W (for BW >=50 kg).
Period: Double-blind Period (up to Week 24)
Arm/Group | Placebo/Alirocumab Q2W | Alirocumab Q2W | Placebo/Alirocumab Q4W | Alirocumab Q4W
Started (Randomized and treated participants.) | 25 | 49 | 27 | 52
Completed | 25 | 45 | 26 | 49
Not Completed | 0 | 4 | 1 | 3
Not completed — Adverse Event | 0 | 0 | 0 | 2
Not completed — Participant moved | 0 | 1 | 0 | 0
Not completed — Life events made continuing too difficult | 0 | 1 | 0 | 0
Not completed — Participant non-compliance to investigational medicinal product (IMP) | 0 | 2 | 0 | 0
Not completed — Other than specified above | 0 | 0 | 1 | 1
Period: Open Label Period (up to Week 104)
Arm/Group | Placebo/Alirocumab Q2W | Alirocumab Q2W | Placebo/Alirocumab Q4W | Alirocumab Q4W
Started (Post completion of DB treatment period, only eligible participants entered OL treatment period.) | 25 | 46 (Of the completed 45 participants of DB Alirocumab Q2W arm, 1 participant did not enter in OL period, and 2 participants discontinued DB period but entered in OL period) | 25 (Of the completed 26 participants of DB period Placebo arm, 1 participant did not enter in OL period.) | 49
Completed | 22 | 43 | 24 | 49
Not Completed | 3 | 3 | 1 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0
Not completed — Participant moved | 1 | 0 | 1 | 0
Not completed — Life events made continuing too difficult | 0 | 1 | 0 | 0
Not completed — Other than specified above | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all randomized participants.
Groups:
- DB Period: Placebo Q2W: Participants received SC injection of placebo (matched to alirocumab) based on their BW (<50 kg or >=50 kg) Q2W for 24 weeks in DB treatment period along with LMT.
- DB Period: Alirocumab Q2W: Participants received SC injection of alirocumab 40 mg (for BW <50 kg) or 75 mg (for BW >=50 kg) Q2W for 24 weeks in DB treatment period along with LMT. Alirocumab dose was up-titrated to 75 mg or 150 mg Q2W from Week 12, when LDL-C level was >=110 mg/dL (2.85 mmol/L) at Week 8.
- DB Period: Placebo Q4W: Participants received SC injection of placebo (matched to alirocumab) based on their BW (<50 kg or >=50 kg) Q4W for 24 weeks in DB treatment period along with LMT.
- DB Period: Alirocumab Q4W: Participants received SC injection of alirocumab 150 mg (for BW <50 kg) or 300 mg (for BW >=50 kg) Q4W for 24 weeks in DB treatment period along with LMT. Alirocumab dose was up-titrated to 75 mg or 150 mg Q2W from Week 12, when LDL-C level >=110 mg/dL (2.85 mmol/L) at Week 8.
Arm/Group | DB Period: Placebo Q2W | DB Period: Alirocumab Q2W | DB Period: Placebo Q4W | DB Period: Alirocumab Q4W | Total Title
Number analyzed (Participants) | 25 | 49 | 27 | 52 | 153
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.2 (2.4) | 12.5 (2.7) | 12.8 (3.0) | 13.1 (3.0) | 12.9 (2.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 30 | 15 | 34 | 87
  Male | 17 | 19 | 12 | 18 | 66
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 4 | 12 | 16
  Asian | 1 | 1 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 1
  Black or African American | 0 | 1 | 1 | 1 | 3
  White | 23 | 42 | 22 | 38 | 125
  More than one race | 1 | 4 | 0 | 0 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Low-Density Lipoprotein Cholesterol (LDL-C) [Mean (Standard Deviation); unit: milligrams/deciliter (mg/dL)] — Calculated LDL-C values were obtained using Friedewald formula: LDL-C = Total cholesterol - High-density lipoprotein cholesterol [HDL-C] - [Triglyceride/5])
  milligrams/deciliter (mg/dL) | 175.29 (50.23) | 169.69 (46.74) | 176.57 (49.01) | 176.79 (53.93) | 174.23 (49.85)

OUTCOME MEASURES:

1. Primary Outcome: DB Period: Percent Change From Baseline in Low Density Lipoprotein Cholesterol (LDL-C) at Week 24: Intent-to-treat (ITT) Estimand
Description: Adjusted least square (LS) means and standard errors (SE) were obtained from mixed-effect model with repeated measures (MMRM) model. All post-baseline data available up to Week 24 were used and missing data were accounted for by the MMRM model. MMRM model was run on participants with a Baseline value and a post-baseline value for at least one timepoint used in the model.
Time Frame: Baseline, Week 24
Population: Analysis was performed on ITT population which included all randomized participants who were analyzed according to the treatment group allocated by randomization. Here, overall number of participants analyzed = participants with available data for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: percent change
Groups:
- DB Period: Alirocumab Q2W: Participants received SC injection of alirocumab 40 mg (for BW <50 kg) or 75 mg (for BW >=50 kg) Q2W for 24 weeks in DB treatment period along with LMT. Alirocumab dose was up-titrated to 75 mg or 150 mg Q2W from Week 12, when LDL-C level >=110 mg/dL (2.85 mmol/L) at Week 8.
Arm/Group | DB Period: Placebo Q2W | DB Period: Alirocumab Q2W | DB Period: Placebo Q4W | DB Period: Alirocumab Q4W
Number analyzed (Participants) | 25 | 49 | 26 | 50
percent change | 9.7 (4.3) | -33.6 (3.4) | -4.4 (3.7) | -38.2 (4.0)
Statistical Analysis 1: Comparison: DB Period: Placebo Q2W vs DB Period: Alirocumab Q2W; The MMRM model included fixed categorical effects of treatment group (alirocumab, placebo), randomization strata (previous participation [yes or no] to DFI14223 study, Baseline BW [<50 or >=50 kg]) as per interactive voice response system (IVRS), time point, treatment-by-time point interaction, strata-by-time point interaction, as well as the continuous fixed covariates of Baseline LDL-C value and Baseline value by time-point interaction. Comparison was performed using an appropriate contrast; Test type: Superiority — Bonferroni adjustment was applied to handle multiplicity for the comparison of each alirocumab dosing regimen group versus its placebo group for the primary efficacy endpoint; p < 0.0001, MMRM — The threshold for statistical significance was 0.025 level; LS mean difference = -43.3, 97.5% CI 2-sided [-56.0 to -30.7], Standard Error of Mean 5.5 — Alirocumab Q2W versus Placebo Q2W
Statistical Analysis 2: Comparison: DB Period: Placebo Q4W vs DB Period: Alirocumab Q4W; The MMRM model included the fixed categorical effects of treatment group (alirocumab, placebo), randomization strata (Baseline BW [<50 or >=50 kg]) as per IVRS, time point, treatment-by-time point interaction, and BW strata-by-time point interaction, as well as the continuous fixed covariates of Baseline LDL-C value and Baseline value by time-point interaction. Comparison was performed using an appropriate contrast; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, MMRM — The threshold for statistical significance was 0.025 level; LS mean difference = -33.8, 97.5% CI 2-sided [-46.4 to -21.2], Standard Error of Mean 5.5 — Alirocumab Q4W versus Placebo Q4W

2. Secondary Outcome: DB Period: Percent Change From Baseline in Low Density Lipoprotein Cholesterol at Week 12: ITT Estimand
Description: Adjusted LS means and SE were obtained from MMRM model including all available post-baseline data. All post-baseline data available up to Week 12 were used and missing data were accounted for by the MMRM model. MMRM model was run on participants with a Baseline value and a post-baseline value for at least one timepoint used in the model.
Time Frame: Baseline, Week 12
Population: Analysis was performed on ITT population. Here, overall number of participants analyzed = participants with available data for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | DB Period: Placebo Q2W | DB Period: Alirocumab Q2W | DB Period: Placebo Q4W | DB Period: Alirocumab Q4W
Number analyzed (Participants) | 25 | 49 | 26 | 50
percent change | 10.7 (3.6) | -34.8 (3.0) | 2.3 (3.6) | -39.2 (3.3)
Statistical Analysis 1: Comparison: DB Period: Placebo Q2W vs DB Period: Alirocumab Q2W; The MMRM model included the fixed categorical effects of treatment group (alirocumab, placebo), randomization strata (previous participation [yes or no] to DFI14223 study, Baseline BW [<50 or >=50 kg]) as per IVRS, time point, treatment-by-time point interaction, strata-by-time point interaction, as well as the continuous fixed covariates of Baseline LDL-C value and Baseline value by time-point interaction. Comparison was performed using an appropriate contrast; Test type: Superiority — Hierarchical testing method was used to control type I error and handle multiple secondary endpoint analyses. Testing was then performed sequentially in the order the endpoints were reported and independently for each dosing regimen. The hierarchical testing sequence continued only when previous endpoint was statistically significant at 0.025 level. Statistical significance of the primary endpoint was required before testing the first secondary endpoint for each dosing regimen independently; p < 0.0001, MMRM — Threshold for significance at 0.025 level; LS mean difference = -45.5, 97.5% CI 2-sided [-56.3 to -34.7], Standard Error of Mean 4.7 — Alirocumab Q2W versus Placebo Q2W
Statistical Analysis 2: Comparison: DB Period: Placebo Q4W vs DB Period: Alirocumab Q4W; [analysis description as in outcome 1, analysis 2]; Test type: Superiority — A hierarchical testing method was used to control type I error and handle multiple secondary endpoint analyses. Testing was then performed sequentially in the order the endpoints are reported and independently for each dosing regimen. The hierarchical testing sequence continued only when previous endpoint was statistically significant at 0.025 level. Statistical significance of the primary endpoint was required before testing the first secondary endpoint for each dosing regimen independently; p < 0.0001, MMRM — Threshold for significance at 0.025 level; LS mean difference = -41.5, 97.5% CI 2-sided [-52.7 to -30.2], Standard Error of Mean 4.9 — Alirocumab Q4W versus Placebo Q4W

3. Secondary Outcome: DB Period: Percent Change From Baseline in Apolipoprotein B (Apo B) at Week 24: ITT Estimand
Description: Adjusted LS means and SE were obtained from MMRM model including all available post-baseline data. All post-baseline data available up to Week 24 were used and missing data were accounted for by the MMRM model. MMRM model was run on participants with a Baseline value and a post-baseline value for at least one timepoint used in the model.
Time Frame: Baseline, Week 24
Population: Analysis was performed on ITT population. Here, overall number of participants analyzed = participants with available data for this outcome measure.
  .
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | DB Period: Placebo Q2W | DB Period: Alirocumab Q2W | DB Period: Placebo Q4W | DB Period: Alirocumab Q4W
Number analyzed (Participants) | 25 | 47 | 26 | 49
percent change | 10.4 (2.8) | -27.4 (3.2) | -3.6 (3.9) | -34.3 (2.9)
Statistical Analysis 1: Comparison: DB Period: Placebo Q2W vs DB Period: Alirocumab Q2W; The MMRM model included the fixed categorical effects of treatment group (alirocumab, placebo), randomization strata (previous participation [yes or no] to DFI14223 study, Baseline BW [<50 or >=50 kg]) as per IVRS, time point, treatment-by-time point interaction, strata-by-time point interaction, as well as the continuous fixed covariates of Baseline Apo B value and Baseline Apo B value by time-point interaction. Comparison was performed using an appropriate contrast; Test type: Superiority — Testing according to the hierarchical testing procedure (only performed if the previous endpoint was statistically significant for the considered dosing regimen); p < 0.0001, MMRM — Threshold for significance at 0.025 level; LS mean difference = -37.8, 97.5% CI 2-sided [-47.5 to -28.2], Standard Error of Mean 4.2 — Alirocumab Q2W versus Placebo Q2W
Statistical Analysis 2: Comparison: DB Period: Placebo Q4W vs DB Period: Alirocumab Q4W; The MMRM model included the fixed categorical effects of treatment group (alirocumab, placebo), randomization strata (Baseline BW [<50 or >=50 kg]) as per IVRS, time point, treatment-by-time point interaction, and BW strata-by-time point interaction, as well as the continuous fixed covariates of Baseline Apo B value and Baseline Apo B value by time-point interaction. Comparison was performed using an appropriate contrast; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p < 0.0001, MMRM — Threshold for significance at 0.025 level; LS mean difference = -30.7, 97.5% CI 2-sided [-42.0 to -19.4], Standard Error of Mean 4.9 — Alirocumab Q4W versus Placebo Q4W

4. Secondary Outcome: DB Period: Percent Change From Baseline in Non-High Density Lipoprotein Cholesterol (Non-HDL-C) at Week 24: ITT Estimand
Description: as for outcome 3
Time Frame: Baseline, Week 24
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | DB Period: Placebo Q2W | DB Period: Alirocumab Q2W | DB Period: Placebo Q4W | DB Period: Alirocumab Q4W
Number analyzed (Participants) | 25 | 49 | 26 | 50
percent change | 9.7 (3.9) | -31.0 (3.2) | -3.7 (4.0) | -35.6 (3.5)
Statistical Analysis 1: Comparison: DB Period: Placebo Q2W vs DB Period: Alirocumab Q2W; The MMRM model included the fixed categorical effects of treatment group (alirocumab, placebo), randomization strata (previous participation [yes or no] to DFI14223 study, Baseline BW [<50 or >=50 kg]) as per IVRS, time point, treatment-by-time point interaction, strata-by-time point interaction, as well as the continuous fixed covariates of Baseline non-HDL-C value and Baseline non-HDL-C value by time-point interaction. Comparison was performed using an appropriate contrast; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p < 0.0001, MMRM — Threshold for significance at 0.025 level; LS mean difference = -40.7, 97.5% CI 2-sided [-52.2 to -29.1], Standard Error of Mean 5.0 — Alirocumab Q2W versus Placebo Q2W
Statistical Analysis 2: Comparison: DB Period: Placebo Q4W vs DB Period: Alirocumab Q4W; The MMRM model included the fixed categorical effects of treatment group (alirocumab, placebo), randomization strata (Baseline BW [<50 or >=50 kg]) as per IVRS, time point, treatment-by-time point interaction, and BW strata-by-time point interaction, as well as the continuous fixed covariates of Baseline non-HDL-C value and Baseline non-HDL-C value by time-point interaction. Comparison was performed using an appropriate contrast; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p < 0.0001, MMRM — Threshold for significance at 0.025 level; LS mean difference = -31.9, 97.5% CI 2-sided [-44.1 to -19.7], Standard Error of Mean 5.3 — Alirocumab Q4W versus Placebo Q4W

5. Secondary Outcome: DB Period: Percent Change From Baseline in Total Cholesterol (Total-C) at Week 24: ITT Estimand
Description: as for outcome 3
Time Frame: Baseline, Week 24
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | DB Period: Placebo Q2W | DB Period: Alirocumab Q2W | DB Period: Placebo Q4W | DB Period: Alirocumab Q4W
Number analyzed (Participants) | 25 | 49 | 26 | 50
percent change | 7.4 (3.0) | -23.4 (2.5) | -4.4 (3.3) | -27.7 (2.9)
Statistical Analysis 1: Comparison: DB Period: Placebo Q2W vs DB Period: Alirocumab Q2W; The MMRM model included the fixed categorical effects of treatment group (alirocumab, placebo), randomization strata (previous participation [yes or no] to DFI14223 study, Baseline BW [<50 or >=50 kg]) as per IVRS, time point, treatment-by-time point interaction, strata-by-time point interaction, as well as the continuous fixed covariates of Baseline Total-C value and Baseline Total-C value by time-point interaction. Comparison was performed using an appropriate contrast; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p < 0.0001, MMRM — Threshold for significance at 0.025 level; LS mean difference = -30.8, 97.5% CI 2-sided [-39.8 to -21.9], Standard Error of Mean 3.9 — Alirocumab Q2W versus Placebo Q2W
Statistical Analysis 2: Comparison: DB Period: Placebo Q4W vs DB Period: Alirocumab Q4W; The MMRM model included the fixed categorical effects of treatment group (alirocumab, placebo), randomization strata (Baseline BW [<50 or >=50 kg]) as per IVRS, time point, treatment-by-time point interaction, and BW strata-by-time point interaction, as well as the continuous fixed covariates of Baseline Total-C value and Baseline Total-C value by time-point interaction. Comparison was performed using an appropriate contrast; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p < 0.0001, MMRM — Threshold for significance at 0.025 level; LS mean difference = -23.3, 97.5% CI 2-sided [-33.5 to -13.1], Standard Error of Mean 4.4 — Alirocumab Q4W versus Placebo Q4W

6. Secondary Outcome: DB Period: Percent Change From Baseline in Apolipoprotein B at Week 12: ITT Estimand
Description: as for outcome 2
Time Frame: Baseline, Week 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | DB Period: Placebo Q2W | DB Period: Alirocumab Q2W | DB Period: Placebo Q4W | DB Period: Alirocumab Q4W
Number analyzed (Participants) | 25 | 47 | 26 | 49
percent change | 8.9 (3.1) | -30.0 (2.5) | 1.1 (3.2) | -31.7 (2.9)
Statistical Analysis 1: Comparison: DB Period: Placebo Q2W vs DB Period: Alirocumab Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p < 0.0001, MMRM — Threshold for significance at 0.025 level; LS mean difference = -38.9, 97.5% CI 2-sided [-48.2 to -29.6], Standard Error of Mean 4.0 — Alirocumab Q2W versus Placebo Q2W
Statistical Analysis 2: Comparison: DB Period: Placebo Q4W vs DB Period: Alirocumab Q4W; [analysis description as in outcome 3, analysis 2]; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p < 0.0001, MMRM; LS mean difference = -32.8, 97.5% CI 2-sided [-42.8 to -22.7], Standard Error of Mean 4.3 — Alirocumab Q4W versus Placebo Q4W

7. Secondary Outcome: DB Period: Percent Change From Baseline in Non-High Density Lipoprotein Cholesterol at Week 12: ITT Estimand
Description: as for outcome 2
Time Frame: Baseline, Week 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | DB Period: Placebo Q2W | DB Period: Alirocumab Q2W | DB Period: Placebo Q4W | DB Period: Alirocumab Q4W
Number analyzed (Participants) | 25 | 49 | 26 | 50
percent change | 9.8 (3.8) | -33.0 (2.8) | 2.8 (3.5) | -34.7 (2.9)
Statistical Analysis 1: Comparison: DB Period: Placebo Q2W vs DB Period: Alirocumab Q2W; [analysis description as in outcome 4, analysis 1]; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p < 0.0001, MMRM — Threshold for significance at 0.025 level; LS mean difference = -42.8, 97.5% CI 2-sided [-53.8 to -31.8], Standard Error of Mean 4.7 — Alirocumab Q2W versus Placebo Q2W
Statistical Analysis 2: Comparison: DB Period: Placebo Q4W vs DB Period: Alirocumab Q4W; [analysis description as in outcome 4, analysis 2]; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p < 0.0001, MMRM — Threshold for significance at 0.025 level; LS mean difference = -37.5, 97.5% CI 2-sided [-47.9 to -27.0], Standard Error of Mean 4.5 — Alirocumab Q4W versus Placebo Q4W

8. Secondary Outcome: DB Period: Percent Change From Baseline in Total Cholesterol at Week 12: ITT Estimand
Description: as for outcome 2
Time Frame: Baseline, Week 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | DB Period: Placebo Q2W | DB Period: Alirocumab Q2W | DB Period: Placebo Q4W | DB Period: Alirocumab Q4W
Number analyzed (Participants) | 25 | 49 | 26 | 50
percent change | 7.5 (2.9) | -25.3 (2.2) | 0.9 (2.5) | -27.0 (2.3)
Statistical Analysis 1: Comparison: DB Period: Placebo Q2W vs DB Period: Alirocumab Q2W; [analysis description as in outcome 5, analysis 1]; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p < 0.0001, MMRM — Threshold for significance at 0.025 level; LS mean difference = -32.7, 97.5% CI 2-sided [-41.3 to -24.2], Standard Error of Mean 3.7 — Alirocumab Q2W versus Placebo Q2W
Statistical Analysis 2: Comparison: DB Period: Placebo Q4W vs DB Period: Alirocumab Q4W; [analysis description as in outcome 5, analysis 2]; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p < 0.0001, MMRM — Threshold for significance at 0.025 level; LS mean difference = -27.9, 97.5% CI 2-sided [-35.6 to -20.2], Standard Error of Mean 3.4 — Alirocumab Q4W versus Placebo Q4W

9. Secondary Outcome: DB Period: Percentage of Participants Who Achieved Low Density Lipoprotein Cholesterol Level Lower Than (<) 130 mg/dL (3.37 mmol/L) at Week 24: ITT Estimand
Description: Adjusted percentages at Week 24 were obtained from multiple imputation approach for handling of missing data. All available post-baseline data up to Week 24 were included in the imputation model.
Time Frame: At Week 24
Population: Analysis was performed on ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | DB Period: Placebo Q2W | DB Period: Alirocumab Q2W | DB Period: Placebo Q4W | DB Period: Alirocumab Q4W
Number analyzed (Participants) | 25 | 49 | 27 | 52
percentage of participants | 8.0 | 73.3 | 22.2 | 76.3
Statistical Analysis 1: Comparison: DB Period: Placebo Q2W vs DB Period: Alirocumab Q2W; Multiple imputation approach followed by logistic regression model. Logistic regression model stratified by randomization factors (previous participation [yes or no] to DFI14223 study, Baseline BW [<50 or >=50 kg]) as per IVRS included the fixed categorical effect of treatment group and the continuous fixed covariate of Baseline LDL-C value; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.0001, Regression, Logistic — Threshold for significance at 0.025 level; Odds Ratio (OR) = 77.6, 97.5% CI 2-sided [6.3 to 960.0] — Alirocumab Q2W versus Placebo Q2W: Combined estimate for odds ratio was obtained by combining the logarithm of odds ratio from logistic regression model analyses of the different imputed data sets, using Rubin's formulae
Statistical Analysis 2: Comparison: DB Period: Placebo Q4W vs DB Period: Alirocumab Q4W; Multiple imputation approach followed by logistic regression model. Logistic regression model stratified by randomization factors (Baseline BW [<50 or >=50 kg]) as per IVRS included the fixed categorical effect of treatment group and the continuous fixed covariate of Baseline LDL-C value; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p < 0.0001, Regression, Logistic — Threshold for significance at 0.025 level; Odds Ratio (OR) = 14.9, 97.5% CI 2-sided [3.2 to 69.8] — Alirocumab Q4W versus Placebo Q4W: Combined estimate for odds ratio was obtained by combining the logarithm of odds ratio from logistic regression model analyses of the different imputed data sets, using Rubin's formulae

10. Secondary Outcome: DB Period: Percentage of Participants Who Achieved Low Density Lipoprotein Cholesterol Level <130 mg/dL (3.37 mmol/L) at Week 12: ITT Estimand
Description: Adjusted percentages at Week 12 were obtained from multiple imputation approach for handling of missing data. All available post-baseline data up to Week 12 were included in the imputation model.
Time Frame: At Week 12
Population: Analysis was performed on ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | DB Period: Placebo Q2W | DB Period: Alirocumab Q2W | DB Period: Placebo Q4W | DB Period: Alirocumab Q4W
Number analyzed (Participants) | 25 | 49 | 27 | 52
percentage of participants | 16.4 | 70.6 | 12.9 | 72.6
Statistical Analysis 1: Comparison: DB Period: Placebo Q2W vs DB Period: Alirocumab Q2W; Multiple imputation approach followed by logistic regression model. The logistic regression model stratified by randomization factors (previous participation [yes or no] to DFI14223 study, Baseline BW [<50 or >=50 kg]) as per IVRS included the fixed categorical effect of treatment group and the continuous fixed covariate of Baseline LDL-C value; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p < 0.0001, Regression, Logistic — Threshold for significance at 0.025 level; Odds Ratio (OR) = 26.5, 97.5% CI 2-sided [4.0 to 174.8] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 2: Comparison: DB Period: Placebo Q4W vs DB Period: Alirocumab Q4W; Multiple imputation approach followed by logistic regression model. The logistic regression model stratified by randomization factors (Baseline BW [<50 or >=50 kg]) as per IVRS included the fixed categorical effect of treatment group and the continuous fixed covariate of Baseline LDL-C value; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p < 0.0001, Regression, Logistic — Threshold for significance at 0.025 level; Odds Ratio (OR) = 40.9, 97.5% CI 2-sided [5.7 to 290.9] — [estimate comment as in outcome 9, analysis 2]

11. Secondary Outcome: DB Period: Percentage of Participants Achieving Low Density Lipoprotein Cholesterol <110 mg/dL (2.84 mmol/L) at Week 24: ITT Estimand
Description: as for outcome 9
Time Frame: At Week 24
Population: Analysis was performed on ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | DB Period: Placebo Q2W | DB Period: Alirocumab Q2W | DB Period: Placebo Q4W | DB Period: Alirocumab Q4W
Number analyzed (Participants) | 25 | 49 | 27 | 52
percentage of participants | 4.0 | 57.2 | 9.0 | 67.2
Statistical Analysis 1: Comparison: DB Period: Placebo Q2W vs DB Period: Alirocumab Q2W; [analysis description as in outcome 10, analysis 1]; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.0011, Regression, Logistic — Threshold for significance at 0.025 level; Odds Ratio (OR) = 52.7, 97.5% CI 2-sided [3.5 to 804.3] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 2: Comparison: DB Period: Placebo Q4W vs DB Period: Alirocumab Q4W; [analysis description as in outcome 10, analysis 2]; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.0006, Regression, Logistic — Threshold for significance at 0.025 level; Odds Ratio (OR) = 43.1, 97.5% CI 2-sided [3.7 to 498.6] — [estimate comment as in outcome 9, analysis 2]

12. Secondary Outcome: DB Period: Percentage of Participants Achieving Low Density Lipoprotein Cholesterol <110 mg/dL (2.84 mmol/L) at Week 12: ITT Estimand
Description: Adjusted percentages at Week 12 were obtained from multiple imputation approach for handling of missing data for Q4W. All available post-baseline data up to Week 12 were included in the imputation model. For Q2W, adjusted percentages at Week 12 were obtained from last observation carried forward approach (LOCF) to handle missing on-treatment LDL-C values as well as missing post-treatment LDL-C values in participants who discontinued treatment due to the coronavirus disease-2019 pandemic. Other post-treatment missing values were considered as failure.
Time Frame: At Week 12
Population: Analysis was performed on ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | DB Period: Placebo Q2W | DB Period: Alirocumab Q2W | DB Period: Placebo Q4W | DB Period: Alirocumab Q4W
Number analyzed (Participants) | 25 | 49 | 27 | 52
percentage of participants | 0.0 | 61.2 | 4.3 | 57.0
Statistical Analysis 1: Comparison: DB Period: Placebo Q2W vs DB Period: Alirocumab Q2W; The LOCF approach followed by exact conditional logistic regression model. The exact conditional logistic regression model stratified by randomization factors (previous participation [yes or no] to DFI14223 study, Baseline BW [<50 or >=50 kg]) as per IVRS included the fixed categorical effect of treatment group and the quartiles of the Baseline LDL-C value; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p < 0.0001, Exact conditional logistic regression — Threshold for significance at 0.025 level; Odds Ratio (OR) = 41.3, 97.5% CI 2-sided [lower limit 6.6] (The percentage of participants reaching LDL-C level lower than 110 mg/dL was 0% in the placebo arm, as a result it was possible to derive the estimated odds-ratio, but the estimated confidence interval (CI) was very wide, with the upper limit estimated to Infinity, therefore upper limit of 97.5% CI was not available to report.) — Alirocumab Q2W versus Placebo Q2W: Odds ratios and confidence intervals estimated from exact conditional logistic regression model
Statistical Analysis 2: Comparison: DB Period: Placebo Q4W vs DB Period: Alirocumab Q4W; [analysis description as in outcome 10, analysis 2]; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.0005, Regression, Logistic — Threshold for significance at 0.025 level; Odds Ratio (OR) = 104.8, 97.5% CI 2-sided [5.2 to 2095.9] — [estimate comment as in outcome 9, analysis 2]

13. Secondary Outcome: DB Period: Percent Change From Baseline in Lipoprotein (a) at Week 24: ITT Estimand
Description: Adjusted means and standard errors were obtained from a multiple imputation approach followed by a robust regression model including all available post-baseline data up to Week 24. Combined estimates and SE were obtained by combining adjusted means and SE from robust regression model analyses of the different imputed data sets.
Time Frame: Baseline, Week 24
Population: Analysis was performed on ITT population.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | DB Period: Placebo Q2W | DB Period: Alirocumab Q2W | DB Period: Placebo Q4W | DB Period: Alirocumab Q4W
Number analyzed (Participants) | 25 | 49 | 27 | 52
percent change | 0.5 (5.3) | -14.7 (4.1) | 2.5 (7.1) | -22.4 (5.0)
Statistical Analysis 1: Comparison: DB Period: Placebo Q2W vs DB Period: Alirocumab Q2W; Multiple imputation approach followed by robust regression model. The robust regression model included the fixed categorical effect of treatment group and randomization strata (previous participation [yes or no] to DFI14223 study, Baseline BW [<50 or >=50 kg]) as per IVRS and the continuous fixed covariate of Baseline lipoprotein (a) value; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.0237, Robust regression model — Threshold for significance at 0.025 level; Adjusted mean difference = -15.2, 97.5% CI 2-sided [-30.3 to -0.1], Standard Error of Mean 6.7 — Alirocumab Q2W versus Placebo Q2W
Statistical Analysis 2: Comparison: DB Period: Placebo Q4W vs DB Period: Alirocumab Q4W; Multiple imputation approach followed by robust regression model. The robust regression model included the fixed categorical effect of treatment group and randomization strata (Baseline BW [<50 or >=50 kg]) as per IVRS and the continuous fixed covariate of Baseline lipoprotein (a) value; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.0043, Robust regression model — Threshold for significance at 0.025 level; Adjusted mean difference = -24.9, 97.5% CI 2-sided [-44.4 to -5.4], Standard Error of Mean 8.7 — Alirocumab Q4W versus Placebo Q4W

14. Secondary Outcome: DB Period: Percent Change From Baseline in Lipoprotein (a) at Week 12: ITT Estimand
Description: Adjusted means and standard errors were obtained from a multiple imputation approach followed by a robust regression model including all available post-baseline data up to Week 12. Combined estimates and SE were obtained by combining adjusted means and SE from robust regression model analyses of the different imputed data sets.
Time Frame: Baseline, Week 12
Population: Analysis was performed on ITT population.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | DB Period: Placebo Q2W | DB Period: Alirocumab Q2W | DB Period: Placebo Q4W | DB Period: Alirocumab Q4W
Number analyzed (Participants) | 25 | 49 | 27 | 52
percent change | -7.1 (5.9) | -12.7 (3.9) | -2.5 (6.9) | -16.0 (5.1)
Statistical Analysis 1: Comparison: DB Period: Placebo Q2W vs DB Period: Alirocumab Q2W; [analysis description as in outcome 13, analysis 1]; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.4288, Robust regression model — Threshold for significance at 0.025 level; Adjusted mean difference = -5.6, 97.5% CI 2-sided [-21.7 to 10.4], Standard Error of Mean 7.1 — Alirocumab Q2W versus Placebo Q2W
Statistical Analysis 2: Comparison: DB Period: Placebo Q4W vs DB Period: Alirocumab Q4W; [analysis description as in outcome 13, analysis 2]; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.1148, Robust regression model — Threshold for significance at 0.025 level; Adjusted mean difference = -13.5, 97.5% CI 2-sided [-32.7 to 5.7], Standard Error of Mean 8.6 — Alirocumab Q4W versus Placebo Q4W

15. Secondary Outcome: DB Period: Percent Change From Baseline in High-Density Lipoprotein Cholesterol (HDL-C) at Week 24: ITT Estimand
Description: Adjusted LS means and SE were obtained from MMRM model. All post-baseline data available up to Week 24 were used and missing data were accounted for by the MMRM model. MMRM model was run on participants with a Baseline value and a post-baseline value for at least one timepoint used in the model.
Time Frame: Baseline, Week 24
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | DB Period: Placebo Q2W | DB Period: Alirocumab Q2W | DB Period: Placebo Q4W | DB Period: Alirocumab Q4W
Number analyzed (Participants) | 25 | 49 | 26 | 50
percent change | -0.8 (2.1) | 5.6 (1.4) | -1.1 (2.7) | 3.4 (2.1)

16. Secondary Outcome: DB Period: Percent Change From Baseline in Fasting Triglycerides (TG) at Week 24: ITT Estimand
Description: as for outcome 13
Time Frame: Baseline, Week 24
Population: Analysis was performed on ITT population.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | DB Period: Placebo Q2W | DB Period: Alirocumab Q2W | DB Period: Placebo Q4W | DB Period: Alirocumab Q4W
Number analyzed (Participants) | 25 | 49 | 27 | 52
percent change | 7.7 (8.4) | 11.9 (6.3) | 12.2 (8.2) | -6.8 (5.5)

17. Secondary Outcome: DB Period: Percent Change From Baseline in Apolipoprotein A1 (Apo A1) at Week 24: ITT Estimand
Description: as for outcome 15
Time Frame: Baseline, Week 24
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | DB Period: Placebo Q2W | DB Period: Alirocumab Q2W | DB Period: Placebo Q4W | DB Period: Alirocumab Q4W
Number analyzed (Participants) | 25 | 47 | 26 | 49
percent change | -0.1 (2.6) | 1.0 (1.5) | -4.5 (2.6) | 4.4 (2.0)

18. Secondary Outcome: DB Period: Percent Change From Baseline in High-Density Lipoprotein Cholesterol at Week 12: ITT Estimand
Description: Adjusted LS means and SE were obtained from MMRM model. All post-baseline data available up to Week 12 were used and missing data were accounted for by the MMRM model. MMRM model was run on participants with a Baseline value and a post-baseline value for at least one timepoint used in the model.
Time Frame: Baseline, Week 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | DB Period: Placebo Q2W | DB Period: Alirocumab Q2W | DB Period: Placebo Q4W | DB Period: Alirocumab Q4W
Number analyzed (Participants) | 25 | 49 | 26 | 50
percent change | -2.2 (3.2) | 3.5 (2.0) | -3.5 (3.2) | 4.0 (2.2)

19. Secondary Outcome: DB Period: Percent Change From Baseline in Fasting Triglycerides (TG) at Week 12: ITT Estimand
Description: as for outcome 14
Time Frame: Baseline, Week 12
Population: Analysis was performed on ITT population.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | DB Period: Placebo Q2W | DB Period: Alirocumab Q2W | DB Period: Placebo Q4W | Db Period: Alirocumab Q4W
Number analyzed (Participants) | 25 | 49 | 27 | 52
percent change | 6.5 (7.4) | -2.2 (5.0) | 7.8 (8.4) | -0.3 (6.0)

20. Secondary Outcome: DB Period: Percent Change From Baseline in Apolipoprotein A1 at Week 12: ITT Estimand
Description: as for outcome 18
Time Frame: Baseline, Week 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | DB Period: Placebo Q2W | DB Period: Alirocumab Q2W | DB Period: Placebo Q4W | DB Period: Alirocumab Q4W
Number analyzed (Participants) | 25 | 47 | 26 | 49
percent change | -0.1 (1.8) | -1.7 (1.7) | -0.7 (3.1) | 5.0 (1.7)

21. Secondary Outcome: DB Period: Percent Change From Baseline in Low Density Lipoprotein Cholesterol at Weeks 12, and 24: On-treatment Estimand
Description: Adjusted LS means and SE were obtained from MMRM model. All post-baseline on-treatment data available up to Week 12 and Week 24 were used for the MMRM model, i.e., for Q2W data: from 1st investigational medicinal product (IMP) injection up to last IMP injection + 21 days and for Q4W data: from 1st IMP injection up to last IMP injection + 35 days for who stopped IMP before switch to Q2W regimen, + 21 days otherwise. MMRM model was run on participants with a Baseline value and at one on-treatment post-baseline value for a timepoint used in the model.
Time Frame: Baseline, Weeks 12, and 24
Population: Analysis was performed on modified intent-to-treat (mITT) population which included all randomized participants who took at least one dose or part of a dose of the IMP injection. Here, overall number of participants analyzed = participants with available data for this outcome measure.
  .
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | DB Period: Placebo Q2W | DB Period: Alirocumab Q2W | DB Period: Placebo Q4W | DB Period: Alirocumab Q4W
Number analyzed (Participants) | 25 | 49 | 26 | 50
percent change
  Week 12 | 10.7 (3.6) | -34.8 (3.0) | 2.3 (3.6) | -39.2 (3.3)
  Week 24 | 9.7 (4.3) | -33.6 (3.4) | -4.4 (3.7) | -38.2 (4.0)

22. Secondary Outcome: DB Period: Percent Change From Baseline in Apolipoprotein B at Weeks 12 and 24: On-treatment Estimand
Description: Adjusted LS means and SE were obtained from MMRM model. All post-baseline on-treatment data available up to Week 12 and Week 24 were used for the MMRM model, i.e., for Q2W data: from 1st IMP injection up to last IMP injection + 21 days and for Q4W data: from 1st IMP injection up to last IMP injection + 35 days for who stopped IMP before switch to Q2W regimen, + 21 days otherwise. MMRM model was run on participants with a Baseline value and at one on-treatment post-baseline value for a timepoint used in the model.
Time Frame: Baseline, Weeks 12 and 24
Population: Analysis was performed on mITT population. Here, overall number of participants analyzed = participants with available data for this outcome measure.
  .
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | DB Period: Placebo Q2W | DB Period: Alirocumab Q2W | DB Period: Placebo Q4W | DB Period: Alirocumab Q4W
Number analyzed (Participants) | 25 | 47 | 26 | 49
percent change
  Week 12 | 8.9 (3.1) | -30.0 (2.5) | 1.1 (3.2) | -31.7 (2.9)
  Week 24 | 10.4 (2.8) | -27.4 (3.2) | -3.6 (3.9) | -34.3 (2.9)

23. Secondary Outcome: DB Period: Percent Change From Baseline in Non-High Density Lipoprotein Cholesterol at Weeks 12 and 24: On-treatment Estimand
Description: as for outcome 22
Time Frame: Baseline, Weeks 12 and 24
Population: as for outcome 22
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | DB Period: Placebo Q2W | DB Period: Alirocumab Q2W | DB Period: Placebo Q4W | Db Period: Alirocumab Q4W
Number analyzed (Participants) | 25 | 49 | 26 | 50
percent change
  Week 12 | 9.8 (3.8) | -33.0 (2.8) | 2.8 (3.5) | -34.7 (2.9)
  Week 24 | 9.7 (3.9) | -31.0 (3.2) | -3.7 (4.0) | -35.6 (3.5)

24. Secondary Outcome: DB Period: Percent Change From Baseline in Total Cholesterol at Weeks 12 and 24: On-treatment Estimand
Description: as for outcome 22
Time Frame: Baseline, Weeks 12 and 24
Population: as for outcome 22
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | DB Period: Placebo Q2W | DB Period: Alirocumab Q2W | DB Period: Placebo Q4W | DB Period: Alirocumab Q4W
Number analyzed (Participants) | 25 | 49 | 26 | 50
percent change
  Week 12 | 7.5 (2.9) | -25.3 (2.2) | 0.9 (2.5) | -27.0 (2.3)
  Week 24 | 7.4 (3.0) | -23.4 (2.5) | -4.4 (3.3) | -27.7 (2.9)

25. Secondary Outcome: DB Period: Percentage of Participants Who Achieved Low Density Lipoprotein Cholesterol < 130 mg/dL (3.37 mmol/L) at Weeks 12 and 24: On-treatment Estimand
Description: Adjusted percentages at Weeks 12 and 24 were obtained from multiple imputation approach for handling of missing data followed by logistic regression model. All available post-baseline on-treatment data up to Week 12 and Week 24 were included in the imputation model, i.e., for Q2W data: from 1st IMP injection up to last IMP injection + 21 days and for Q4W data: from 1st IMP injection up to last IMP injection + 35 days for those who stopped IMP before switch to Q2W regimen, + 21 days otherwise.
Time Frame: Weeks 12 and 24
Population: Analysis was performed on mITT population.
Measure: Number; unit: percentage of participants
Arm/Group | DB Period: Placebo Q2W | DB Period: Alirocumab Q2W | Db Period: Placebo Q4W | DB Period: Alirocumab Q4W
Number analyzed (Participants) | 25 | 49 | 27 | 52
percentage of participants
  Week 12 | 16.4 | 70.6 | 12.9 | 72.6
  Week 24 | 8.0 | 73.3 | 22.2 | 76.3

26. Secondary Outcome: DB Period: Percentage of Participants Who Achieved Low Density Lipoprotein Cholesterol < 110 mg/dL (2.84 mmol/L) at Weeks 12 and 24: On-treatment Estimand
Description: as for outcome 25
Time Frame: Weeks 12 and 24
Population: Analysis was performed on mITT population.
Measure: Number; unit: percentage of participants
Arm/Group | DB Period: Placebo Q2W | DB Period: Alirocumab Q2W | DB Period: Placebo Q4W | DB Period: Alirocumab Q4W
Number analyzed (Participants) | 25 | 49 | 27 | 52
percentage of participants
  Week 12 | 0.1 | 61.7 | 4.3 | 57.0
  Week 24 | 4.0 | 57.2 | 9.0 | 67.2

27. Secondary Outcome: DB Period: Percent Change From Baseline in Lipoprotein (a) at Weeks 12 and 24: On-treatment Estimand
Description: Adjusted means and standard errors were obtained from a multiple imputation approach followed by a robust regression model including all available post-baseline on-treatment data up to Week 12 and Week 24, i.e., for Q2W data: from 1st IMP injection up to last IMP injection + 21 days and for Q4W data: from 1st IMP injection up to last IMP injection + 35 days for those who stopped IMP before switch to Q2W regimen, + 21 days otherwise. Combined estimates and SE were obtained by combining adjusted means and SE from robust regression model analyses of the different imputed data sets.
Time Frame: Baseline, Weeks 12 and 24
Population: Analysis was performed on mITT population.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | DB Period: Placebo Q2W | DB Period: Alirocumab Q2W | DB Period: Placebo Q4W | DB Period: Alirocumab Q4W
Number analyzed (Participants) | 25 | 49 | 27 | 52
percent change
  Week 12 | -7.099 (5.923) | -12.746 (3.889) | -2.545 (6.851) | -16.042 (5.139)
  Week 24 | 0.492 (5.254) | -14.748 (4.083) | 2.468 (7.135) | -22.418 (5.030)

28. Secondary Outcome: DB Period: Percent Change From Baseline in Apolipoprotein A1 at Weeks 12 and 24: On-treatment Estimand
Description: Adjusted LS means and SE were obtained from MMRM model. All post-baseline on-treatment data available up to Week 12 and Week 24 were used for the MMRM mode, i.e., for Q2W data: from 1st IMP injection up to last IMP injection + 21 days and for Q4W data: from 1st IMP injection up to last IMP injection + 35 days for who stopped IMP before switch to Q2W regimen, + 21 days otherwise. MMRM model was run on participants with a Baseline value and at one on-treatment post-baseline value for a timepoint used in the model.
Time Frame: Baseline, Weeks 12 and 24
Population: as for outcome 22
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | DB Period: Placebo Q2W | DB Period: Alirocumab Q2W | DB Period: Placebo Q4W | DB Period: Alirocumab Q4W
Number analyzed (Participants) | 25 | 47 | 26 | 49
percent change
  Week 12 | -0.1 (1.8) | -1.7 (1.7) | -0.7 (3.1) | 5.0 (1.7)
  Week 24 | -0.1 (2.6) | 1.0 (1.5) | -4.5 (2.6) | 4.4 (2.0)

29. Secondary Outcome: DB Period: Percent Change From Baseline in High-Density Lipoprotein Cholesterol (HDL-C) at Weeks 12 and 24: On-treatment Estimand
Description: Adjusted LS means and SE were obtained from MMRM model. All post-baseline on-treatment data available up to Week 12 and Week 24 were used for the MMRM model, i.e., for Q2W data: from 1st IMP injection up to last IMP injection + 21 days and for Q4W data: from 1st IMP injection up to last IMP injection + 35 days for who stopped IMP before switch to Q2W regimen, + 21 day otherwise. MMRM model was run on participants with a Baseline value and at one on-treatment post-baseline value for a timepoint used in the model.
Time Frame: Baseline, Weeks 12, and 24
Population: as for outcome 22
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | DB Period: Placebo Q2W | DB Period: Alirocumab Q2W | DB Period: Placebo Q4W | DB Period: Alirocumab Q4W
Number analyzed (Participants) | 25 | 49 | 26 | 50
percent change
  Week 12 | -2.2 (3.2) | 3.5 (2.0) | -3.5 (3.2) | 4.0 (2.2)
  Week 24 | -0.8 (2.1) | 5.6 (1.4) | -1.1 (2.7) | 3.4 (2.1)

30. Secondary Outcome: DB Period: Percent Change From Baseline in Fasting Triglycerides at Weeks 12 and 24: On-treatment Estimand
Description: as for outcome 27
Time Frame: Baseline, Weeks 12, and 24
Population: Analysis was performed on mITT population.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | DB Period: Placebo Q2W | DB Period: Alirocumab Q2W | DB Period: Placebo Q4W | DB Period: Alirocumab Q4W
Number analyzed (Participants) | 25 | 49 | 27 | 52
percent change
  Week 12 | 6.5 (7.4) | -2.2 (5.0) | 7.8 (8.4) | -0.3 (6.0)
  Week 24 | 7.7 (8.4) | 11.9 (6.3) | 12.2 (8.2) | -6.8 (5.5)

31. Secondary Outcome: DB Period: Absolute Change From Baseline in Apo B/Apo A-1 Ratio at Weeks 12 and 24: ITT Estimand
Description: Adjusted LS means and SE were obtained from MMRM model. All post-baseline data available up to Week 12 and Week 24 were used and missing data were accounted for by the MMRM model. MMRM model was run on participants with a Baseline value and a post-baseline value for at least one timepoint used in the model.
Time Frame: Baseline, Weeks 12, and 24
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: ratio (Apo B/Apo A-1)
Arm/Group | DB Period: Placebo Q2W | DB Period: Alirocumab Q2W | DB Period: Placebo Q4W | DB Period: Alirocumab Q4W
Number analyzed (Participants) | 25 | 47 | 26 | 49
ratio (Apo B/Apo A-1)
  Week 12 | 0.1 (0.0) | -0.2 (0.0) | 0.0 (0.0) | -0.3 (0.0)
  Week 24 | 0.1 (0.0) | -0.2 (0.0) | 0.0 (0.0) | -0.3 (0.0)

32. Secondary Outcome: DB Period: Absolute Change From Baseline in Apo B/Apo A-1 Ratio at Weeks 12 and 24: On-treatment Estimand
Description: as for outcome 22
Time Frame: Baseline, Weeks 12, and 24
Population: as for outcome 22
Measure: Least Squares Mean (Standard Error); unit: ratio (Apo B/Apo A-1)
Arm/Group | DB Period: Placebo Q2W | DB Period: Alirocumab Q2W | DB Period: Placebo Q4W | DB Period: Alirocumab Q4W
Number analyzed (Participants) | 25 | 47 | 26 | 49
ratio (Apo B/Apo A-1)
  Week 12 | 0.1 (0.0) | -0.2 (0.0) | 0.0 (0.0) | -0.3 (0.0)
  Week 24 | 0.1 (0.0) | -0.2 (0.0) | 0.0 (0.0) | -0.3 (0.0)

33. Secondary Outcome: DB Period: Percentage of Participants Who Achieved at Least 30 Percent (%) Reduction in Low Density Lipoprotein Cholesterol Level From Baseline at Weeks 12 and 24: ITT Estimand
Description: Adjusted percentages at Weeks 12 and 24 were obtained from multiple imputation approach for handling of missing data followed by logistic regression model. All available post-baseline on-treatment data up to Week 12 and Week 24 were included in the imputation model.
Time Frame: At Weeks 12 and 24
Population: Analysis was performed on ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | DB Period: Placebo Q2W | DB Period: Alirocumab Q2W | DB Period: Placebo Q4W | DB Period: Alirocumab Q4W
Number analyzed (Participants) | 25 | 49 | 27 | 52
percentage of participants
  Week12 | 0.8 | 65.8 | 4.2 | 70.8
  Week 24 | 4.0 | 66.7 | 18.5 | 72.5

34. Secondary Outcome: DB Period: Percentage of Participants Achieved at Least 30% Reduction in Low Density Lipoprotein Cholesterol Level From Baseline at Weeks 12 and 24: On-treatment Estimand
Description: as for outcome 25
Time Frame: At Weeks 12 and 24
Population: Analysis was performed on mITT population.
Measure: Number; unit: percentage of participants
Arm/Group | DB Period: Placebo Q2W | DB Period: Alirocumab Q2W | DB Period: Placebo Q4W | DB Period: Alirocumab Q4W
Number analyzed (Participants) | 25 | 49 | 27 | 52
percentage of participants
  Week 12 | 0.8 | 65.8 | 4.2 | 70.8
  Week 24 | 4.0 | 66.7 | 18.5 | 72.5

35. Secondary Outcome: DB Period: Percentage of Participants Who Achieved at Least 50% Reduction in Low Density Lipoprotein Cholesterol Level From Baseline at Weeks 12 and 24: ITT Estimand
Description: as for outcome 33
Time Frame: At Weeks 12 and 24
Population: Analysis was performed on ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | DB Period: Placebo Q2W | DB Period: Alirocumab Q2W | DB Period: Placebo Q4W | DB Period: Alirocumab Q4W
Number analyzed (Participants) | 25 | 49 | 27 | 52
percentage of participants
  Week 12 | 0.0 | 25.2 | 0.1 | 31.9
  Week 24 | 0.0 | 21.6 | 9.1 | 32.4

36. Secondary Outcome: DB Period: Percentage of Participants Who Achieved at Least 50% Reduction in Low Density Lipoprotein Cholesterol Level From Baseline at Weeks 12 and 24: On-treatment Estimand
Description: as for outcome 25
Time Frame: At Weeks 12 and 24
Population: Analysis was performed on mITT population.
Measure: Number; unit: percentage of participants
Arm/Group | DB Period: Placebo Q2W | DB Period: Alirocumab Q2W | DB Period: Placebo Q4W | DB Period: Alirocumab Q4W
Number analyzed (Participants) | 25 | 49 | 27 | 52
percentage of participants
  Week 12 | 0.0 | 25.2 | 0.1 | 31.9
  Week 24 | 0.0 | 21.6 | 9.1 | 32.4

37. Secondary Outcome: DB Period: Percent Change in Low Density Lipoprotein Cholesterol From Baseline to Weeks 8, 12 and 24: ITT Estimand
Description: Adjusted LS means and SE were obtained from MMRM model. All post-baseline data available up to Week 8, Week 12 and Week 24 were used and missing data were accounted for by the MMRM model.
Time Frame: Baseline to Weeks 8, 12 and 24
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | DB Period: Placebo Q2W | DB Period: Alirocumab Q2W | DB Period: Placebo Q4W | DB Period: Alirocumab Q4W
Number analyzed (Participants) | 25 | 49 | 26 | 50
percent change
  Week 8 | 7.1 (4.2) | -35.4 (3.6) | -3.8 (3.5) | -42.0 (2.8)
  Week 12 | 10.7 (3.6) | -34.8 (3.0) | 2.3 (3.6) | -39.2 (3.3)
  Week 24 | 9.7 (4.3) | -33.6 (3.4) | -4.4 (3.7) | -38.2 (4.0)

38. Secondary Outcome: DB Period: Percent Change in Low Density Lipoprotein Cholesterol From Baseline to Weeks 8, 12 and 24: On-treatment Estimand
Description: Adjusted LS means and SE were obtained from MMRM model. All post-baseline on-treatment data available up to Week 8, Week 12 and Week 24 were used for the MMRM model, i.e., for Q2W data: from 1st IMP injection up to last IMP injection + 21 days and for Q4W data: from 1st IMP injection up to last IMP injection + 35 days for who stopped IMP before switch to Q2W regimen, + 21 days otherwise.
Time Frame: Baseline to Weeks 8, 12 and 24
Population: as for outcome 22
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | DB Period: Placebo Q2W | DB Period: Alirocumab Q2W | DB Period: Placebo Q4W | DB Period: Alirocumab Q4W
Number analyzed (Participants) | 25 | 49 | 26 | 50
percent change
  Week 8 | 7.1 (4.2) | -35.4 (3.6) | -3.8 (3.5) | -42.0 (2.8)
  Week 12 | 10.7 (3.6) | -34.8 (3.0) | 2.3 (3.6) | -39.2 (3.3)
  Week 24 | 9.7 (4.3) | -33.6 (3.4) | -4.4 (3.7) | -38.2 (4.0)

39. Secondary Outcome: OL Period: Percent Change in Low Density Lipoprotein Cholesterol From Baseline to Week 104: ITT Estimand
Description: Percent Change in LDL-C from Baseline to Week 104 was reported in this outcome measure.
Time Frame: Baseline, Week 104
Population: Analysis was performed on ITT population. Here, overall number of participants analyzed = participants with available data for this outcome measure. The IIT estimand was analyzed by considering all the post-baseline (including both on- and post-treatment) LDL-C values for the analysis.
  .
Measure: Least Squares Mean (Standard Error); unit: percent change
Groups:
- OL Period: Placebo/Alirocumab Q2W; OL Period: Alirocumab Q2W: After completion of DB treatment period, eligible participants entered into OL treatment period and received alirocumab 40 mg (for BW <50 kg) or 75 mg (for BW >=50 kg) Q2W from Week 24 up to an additional 80 weeks (i.e., up to Week 104) added to stable LMT. After Week 24, dose up-titrated from 40 mg to 75 mg when BW increased from <50 kg to >=50 kg. From Week 32 up to Week 104, based on participant LDL-C value, alirocumab dose was either up-titrated as 40 mg to 75 mg (for BW <50 kg) or 75 mg to 150 mg (for BW >=50 kg) or down titrated as 75 mg to 40 mg (for BW <50 kg) or 150 mg to 75 mg (for BW >=50 kg).
- OL Period: Placebo/Alirocumab Q4W; OL Period: Alirocumab Q4W: After completion of DB treatment period, eligible participants entered into OL treatment period and received alirocumab 150 mg (for BW <50 kg) or 300 mg (for BW >=50 kg) Q4W from Week 24 up to an additional 80 weeks (i.e., up to Week 104) added to stable LMT. After Week 24, dose up-titrated from 150 mg to 300 mg when BW increased from <50 kg to >=50 kg. From Week 32 up to Week 104, based on participant LDL-C value, alirocumab dose was either up-titrated as 150 mg Q4W to 75 mg Q2W (for BW <50 kg) or 300 mg Q4W to 150 mg Q2W (for BW >=50 kg) or down titrated as 75 mg Q2W to 40 mg Q2W (for BW <50 kg) or 150 mg Q2W to 75 mg Q2W (for BW >=50 kg).
Arm/Group | OL Period: Placebo/Alirocumab Q2W | OL Period: Alirocumab Q2W | OL Period: Placebo/Alirocumab Q4W | OL Period: Alirocumab Q4W
Number analyzed (Participants) | 25 | 45 | 23 | 47
percent change | -23.3 (4.9) | -22.2 (5.6) | -27.1 (7.0) | -23.7 (4.2)

40. Secondary Outcome: OL Period: Percent Change in Low Density Lipoprotein Cholesterol From Baseline to Week 104: On-treatment Estimand
Description: Percent Change in LDL-C from Baseline to Week 104 was reported in this outcome measure.
Time Frame: Baseline, Week 104
Population: Analysis was performed on mITT population. Here, 'overall number of participants analyzed' = participants with available data for this outcome measure. The on-treatment estimand was analyzed using the same imputation model as ITT Estimand, but considered the 'on-treatment' LDL-C values alone for the analysis.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | OL Period: Placebo/Alirocumab Q2W | OL Period: Alirocumab Q2W | OL Period: Placebo/Alirocumab Q4W | OL Period: Alirocumab Q4W
Number analyzed (Participants) | 25 | 45 | 23 | 47
percent change | -22.8 (5.1) | -25.8 (4.9) | -27.6 (7.6) | -23.4 (4.7)

41. Secondary Outcome: Change From Baseline in Cogstate Battery Test - Overall Composite Score at Weeks 24, 68 and 104
Description: Cogstate battery test (cognitive testing system) consisted of detection test (DET), identification test (IDN), one card learning test (OCL) and Groton maze learning test (GML) to assess processing speed, attention, visual learning and executive functioning, respectively. For each test, Z-scores were computed based on participant's age at Baseline and Weeks 24, 68 and 104. Composite score: calculated as mean of Z-scores equally weighted, provided that at least 3 of 4 tests were available and if all of these domains were covered as: attention, through either DET or IDN, visual learning, through OCL and executive function, through GML. There is not minimum/maximum since values were reported as z-score but z-score of 0 means result equals to mean with negative numbers indicating values lower than mean and positive values higher. Positive change in z-score = an improvement in cognition, i.e., a better outcome; and negative change in z-score = worsening in cognition, i.e., a worse outcome.
Time Frame: Baseline, Weeks 24, 68 and 104
Population: Analysis was performed on safety population which consisted of the randomized population who had actually received at least one dose or partial dose of IMP. Here, number analyzed = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: Z-score
Groups:
- Placebo/Alirocumab Q2W: Participants received SC injection of placebo (matched to alirocumab) based on their BW (<50 kg or >=50 kg) Q2W for 24 weeks in DB treatment period added to stable LMT. After completion of DB treatment period, eligible participants entered into OL treatment period and received alirocumab 40 mg (for BW <50 kg) or 75 mg (for BW >=50 kg) Q2W from Week 24 up to an additional 80 weeks (i.e., up to Week 104) added to stable LMT. After Week 24, dose up-titrated from 40 mg to 75 mg when BW increased from <50 kg to >=50 kg. From Week 32 up to Week 104, based on participant LDL-C value, alirocumab dose was either up-titrated as 40 mg to 75 mg (for BW <50 kg) or 75 mg to 150 mg (for BW >=50 kg) or down titrated as 75 mg to 40 mg (for BW <50 kg) or 150 mg to 75 mg (for BW >=50 kg).
- Alirocumab Q2W: Participants received SC injection of alirocumab 40 mg (for BW <50 kg) or 75 mg (for BW >=50 kg) Q2W for 24 weeks in DB treatment period added to stable LMT. Alirocumab dose was up-titrated to 75 mg or 150 mg Q2W from Week 12, when LDL-C level was >=110 mg/dL (2.85 mmol/L) at Week 8. After completion of DB treatment period, eligible participants entered into OL treatment period and received alirocumab 40 mg (for BW <50 kg) or 75 mg (for BW >=50 kg) from Week 24 up to an additional 80 weeks (i.e., up to Week 104) added to stable LMT. After Week 24, dose up-titrated from 40 mg to 75 mg when BW increased from <50 kg to >=50 kg. From Week 32 up to Week 104, based on participant LDL-C value, alirocumab dose was either up-titrated as 40 mg to 75 mg (for BW <50 kg) or 75 mg to 150 mg (for BW >=50 kg) or down titrated as 75 mg to 40 mg (for BW <50 kg) or 150 mg to 75 mg (for BW >=50 kg).
- Placebo/Alirocumab Q4W: Participants received SC injection of placebo (matched to alirocumab) based on their BW (<50 kg or >=50 kg) Q4W for 24 weeks in DB treatment period added to stable LMT. After completion of DB treatment period, eligible participants entered into OL treatment period and received alirocumab 150 mg (for BW <50 kg) or 300 mg (for BW >=50 kg) Q2W from Week 24 up to an additional 80 weeks (i.e., up to Week 104) added to stable LMT. After Week 24, dose up-titrated from 150 mg to 300 mg when BW increased from <50 kg to >=50 kg. From Week 32 up to Week 104, based on participant LDL-C value, alirocumab dose was either up-titrated as 150 mg Q4W to 75 mg Q2W (for BW <50 kg) or 300 mg Q4W to 150 mg Q2W (for BW >=50 kg) or down titrated as 75 mg Q2W to 40 mg Q2W (for BW <50 kg) or 150 mg Q2W to 75 mg Q2W (for BW >=50 kg).
Arm/Group | Placebo/Alirocumab Q2W | Alirocumab Q2W | Placebo/Alirocumab Q4W | Alirocumab Q4W
Number analyzed (Participants) | 25 | 49 | 27 | 52
Z-score
  Week 24: number analyzed (Participants) | 16 | 24 | 16 | 29
  Week 24 | -0.403 (1.008) | -0.313 (0.444) | -0.218 (0.501) | -0.136 (0.637)
  Week 68: number analyzed (Participants) | 13 | 23 | 16 | 28
  Week 68 | -0.421 (1.752) | -0.334 (0.912) | -0.272 (0.814) | -0.263 (0.717)
  Week 104: number analyzed (Participants) | 13 | 21 | 15 | 22
  Week 104 | -0.601 (1.612) | -0.439 (0.917) | -0.393 (0.764) | -0.638 (0.791)

42. Secondary Outcome: Number of Participants With Tanner Staging at Baseline and Weeks 24, 68 and 104
Description: Tanner stage defines physical measurements of development in children and adolescent based on external primary and secondary sex characteristics. Participants were evaluated for pubic hair distribution, breast development (only females) and genital development (only males) and classified in 3 categories as: Prepubescent (defined as a person just before start of the development of adult sexual characteristics), Pubescent (defined as a person at or approaching the age of puberty), Postpubescent (sexually mature or a person who has completed puberty).
Time Frame: Baseline, Weeks 24, 68 and 104
Population: Analysis was performed on safety population. Here, number analyzed = participants with available data for each specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo/Alirocumab Q2W | Alirocumab Q2W | Placebo/Alirocumab Q4W | Alirocumab Q4W
Number analyzed (Participants) | 25 | 49 | 27 | 52
Participants
  Baseline: Boys - Prepubescent: number analyzed (Participants) | 17 | 19 | 12 | 18
  Baseline: Boys - Prepubescent | 1 | 4 | 5 | 0
  Baseline: Boys - Pubescent: number analyzed (Participants) | 17 | 19 | 12 | 18
  Baseline: Boys - Pubescent | 13 | 13 | 4 | 14
  Baseline: Boys - Postpubescent: number analyzed (Participants) | 17 | 19 | 12 | 18
  Baseline: Boys - Postpubescent | 3 | 2 | 3 | 4
  Baseline: Girls - Prepubescent: number analyzed (Participants) | 8 | 30 | 15 | 34
  Baseline: Girls - Prepubescent | 1 | 4 | 1 | 7
  Baseline: Girls - Pubescent: number analyzed (Participants) | 8 | 30 | 15 | 34
  Baseline: Girls - Pubescent | 6 | 16 | 8 | 13
  Baseline: Girls - Postpubescent: number analyzed (Participants) | 8 | 30 | 15 | 34
  Baseline: Girls - Postpubescent | 1 | 10 | 6 | 14
  Week 24: Boys - Prepubescent: number analyzed (Participants) | 17 | 17 | 11 | 17
  Week 24: Boys - Prepubescent | 0 | 3 | 1 | 0
  Week 24: Boys - Pubescent: number analyzed (Participants) | 17 | 17 | 11 | 17
  Week 24: Boys - Pubescent | 13 | 11 | 7 | 12
  Week 24: Boys - Postpubescent: number analyzed (Participants) | 17 | 17 | 11 | 17
  Week 24: Boys - Postpubescent | 4 | 3 | 3 | 5
  Week 24: Girls - Prepubescent: number analyzed (Participants) | 8 | 28 | 12 | 27
  Week 24: Girls - Prepubescent | 1 | 4 | 1 | 2
  Week 24: Girls - Pubescent: number analyzed (Participants) | 8 | 28 | 12 | 27
  Week 24: Girls - Pubescent | 5 | 15 | 6 | 16
  Week 24: Girls - Postpubescent: number analyzed (Participants) | 8 | 28 | 12 | 27
  Week 24: Girls - Postpubescent | 2 | 9 | 5 | 9
  Week 68: Boys - Prepubescent: number analyzed (Participants) | 11 | 16 | 9 | 15
  Week 68: Boys - Prepubescent | 0 | 1 | 1 | 0
  Week 68: Boys - Pubescent: number analyzed (Participants) | 11 | 16 | 9 | 15
  Week 68: Boys - Pubescent | 7 | 9 | 5 | 9
  Week 68: Boys - Postpubescent: number analyzed (Participants) | 11 | 16 | 9 | 15
  Week 68: Boys - Postpubescent | 4 | 6 | 3 | 6
  Week 68: Girls - Prepubescent: number analyzed (Participants) | 7 | 26 | 11 | 26
  Week 68: Girls - Prepubescent | 0 | 3 | 1 | 1
  Week 68: Girls - Pubescent: number analyzed (Participants) | 7 | 26 | 11 | 26
  Week 68: Girls - Pubescent | 6 | 14 | 5 | 16
  Week 68: Girls - Postpubescent: number analyzed (Participants) | 7 | 26 | 11 | 26
  Week 68: Girls - Postpubescent | 1 | 9 | 5 | 9
  Week 104: Boys - Prepubescent: number analyzed (Participants) | 13 | 15 | 8 | 15
  Week 104: Boys - Prepubescent | 0 | 1 | 1 | 0
  Week 104: Boys - Pubescent: number analyzed (Participants) | 13 | 15 | 8 | 15
  Week 104: Boys - Pubescent | 6 | 8 | 5 | 8
  Week 104: Boys - Postpubescent: number analyzed (Participants) | 13 | 15 | 8 | 15
  Week 104: Boys - Postpubescent | 7 | 6 | 2 | 7
  Week 104: Girls - Prepubescent: number analyzed (Participants) | 6 | 21 | 11 | 29
  Week 104: Girls - Prepubescent | 0 | 0 | 1 | 1
  Week 104: Girls - Pubescent: number analyzed (Participants) | 6 | 21 | 11 | 29
  Week 104: Girls - Pubescent | 4 | 10 | 5 | 17
  Week 104: Girls - Postpubescent: number analyzed (Participants) | 6 | 21 | 11 | 29
  Week 104: Girls - Postpubescent | 2 | 11 | 5 | 11

43. Secondary Outcome: DB Period: Number of Participants With Treatment-Emergent (TE) Positive Anti-Alirocumab Antibodies (ADA) Response
Description: Anti-drug (alirocumab) antibodies samples were analyzed using a validated non-quantitative, titer-based bridging immunoassay. Number of participants with positive ADA during 24-week treatment period is reported. Treatment-emergent positive ADA response was defined as 1) participants with no ADA positive response at baseline but with any positive response in the post-baseline period or 2) participants with a positive ADA response at baseline and at least a 4- fold increase in titer in the post-baseline period. A persistent positive response was defined as a TE ADA positive response detected in at least 2 consecutive post-baseline samples separated by at least a 12-week period. Persistent positive response was only analyzed for participants with positive TE ADA response.
Time Frame: Up to 24 weeks
Population: Analysis was performed on ADA population which included all randomized and treated (who actually received at least one dose or part of a dose of the IMP injection) participants with an available ADA sample at Baseline (Week 0) and at least 1 non-missing ADA sample post first IMP injection and up to Week 24/early termination. Here, 'number analyzed' = participants with available data for each specified category and '0' in number analyzed filed signifies that no participants were evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | DB Period: Placebo Q2W | DB Period: Alirocumab Q2W | DB Period: Placebo Q4W | DB Period: Alirocumab Q4W
Number analyzed (Participants) | 25 | 48 | 26 | 49
Participants
  TE ADA positive response | 0 | 3 | 0 | 0
  Persistent positive response: number analyzed (Participants) | 0 | 3 | 0 | 0
  Persistent positive response |  | 0 |  |

ADVERSE EVENTS:
Time Frame: For the DB period: for participants proceeding into the OL treatment period, from first DB IMP dose up to the day before first OL IMP dose ( i.e., up to Week 24); and for participants not proceeding into the OL treatment period, from first DB IMP dose up to Week 24 + 10 weeks (i.e., up to Week 34); for the OL period: from first OL IMP dose up to 10 weeks after the last OL IMP dose (i.e., up to Week 112)
Description: Reported AEs were AEs which developed, worsened/became serious in each of the study periods, i.e. DB and OL, respectively.
Groups:
- OL Period: Alirocumab Q2W: After completion of DB treatment period, eligible participants entered into OL treatment period and received alirocumab 40 mg (for BW <50 kg) or 75 mg (for BW >=50 kg) from Week 24 up to an additional 80 weeks (i.e., up to Week 104) added to stable LMT. After Week 24, dose up-titrated from 40 mg to 75 mg when BW increased from <50 kg to >=50 kg. From Week 32 up to Week 104, based on participant LDL-C value, alirocumab dose was either up-titrated as 40 mg to 75 mg (for BW <50 kg) or 75 mg to 150 mg (for BW >=50 kg) or down titrated as 75 mg to 40 mg (for BW <50 kg) or 150 mg to 75 mg (for BW >=50 kg).
Arm/Group | DB Period: Placebo Q2W | DB Period: Alirocumab Q2W | DB Period: Placebo Q4W | DB Period: Alirocumab Q4W | OL Period: Placebo/Alirocumab Q2W | OL Period: Alirocumab Q2W | OL Period: Placebo/Alirocumab Q4W | OL Period: Alirocumab Q4W
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/49 | 0/27 | 0/52 | 0/25 | 0/46 | 0/25 | 0/49
Serious Adverse Events (participants affected / at risk) | 1/25 | 4/49 | 1/27 | 2/52 | 0/25 | 4/46 | 2/25 | 3/49
Other Adverse Events (participants affected / at risk) | 9/25 | 15/49 | 8/27 | 10/52 | 9/25 | 12/46 | 6/25 | 15/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DB Period: Placebo Q2W (N=25) | DB Period: Alirocumab Q2W (N=49) | DB Period: Placebo Q4W (N=27) | DB Period: Alirocumab Q4W (N=52) | OL Period: Placebo/Alirocumab Q2W (N=25) | OL Period: Alirocumab Q2W (N=46) | OL Period: Placebo/Alirocumab Q4W (N=25) | OL Period: Alirocumab Q4W (N=49)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis Streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Major Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Angina Pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal Hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sympathetic Posterior Cervical Syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Calculus Urinary (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament Rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DB Period: Placebo Q2W (N=25) | DB Period: Alirocumab Q2W (N=49) | DB Period: Placebo Q4W (N=27) | DB Period: Alirocumab Q4W (N=52) | OL Period: Placebo/Alirocumab Q2W (N=25) | OL Period: Alirocumab Q2W (N=46) | OL Period: Placebo/Alirocumab Q4W (N=25) | OL Period: Alirocumab Q4W (N=49)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (5)
Nasopharyngitis (Infections and infestations) | 2 (2) | 7 (7) | 2 (2) | 1 (4) | 2 (2) | 3 (5) | 1 (2) | 3 (5)
Tonsillitis (Infections and infestations) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 3 (3) | 3 (3) | 3 (3) | 3 (3) | 2 (2) | 2 (4) | 0 (0) | 2 (3)
Headache (Nervous system disorders) | 2 (2) | 3 (3) | 1 (1) | 4 (5) | 1 (6) | 5 (5) | 4 (5) | 7 (15)
Migraine (Nervous system disorders) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (2)
Injection Site Reaction (General disorders) | 0 (0) | 3 (12) | 0 (0) | 2 (3) | 1 (2) | 3 (17) | 1 (2) | 1 (1)
Low Density Lipoprotein Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2021-01-06): https://cdn.clinicaltrials.gov/large-docs/84/NCT03510884/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-19): https://cdn.clinicaltrials.gov/large-docs/84/NCT03510884/SAP_001.pdf